CLINICAL TRIAL: NCT00427713
Title: Chemotherapy or No Chemotherapy in Clear Margins After Neoadjuvant Chemoradiation in Locally Advanced Rectal Cancer. A Randomised Phase III Trial of Control Vs Capecitabine Plus Oxaliplatin [CHRONICLE]
Brief Title: Capecitabine and Oxaliplatin or Standard Follow-Up Care in Treating Patients Who Have Undergone Surgery for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000526299; CRUK-CHRONICLE; CRUK-BRD/05/132; EU-20679; ISRCTN59865116; CTA21106/0016/001; EUDRACT-2004-001484-21
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-06

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage III rectal cancer; stage II rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin
Procedure: adjuvant therapy
Procedure: standard follow-up care

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving capecitabine together with oxaliplatin is more effective than standard follow-up care in treating rectal cancer that was removed by surgery.

PURPOSE: This randomized phase III trial is studying capecitabine and oxaliplatin to see how well they work compared with standard follow-up care in treating patients who have undergone surgery for locally advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of adjuvant chemotherapy comprising capecitabine and oxaliplatin vs standard follow-up care, in terms of disease-free and overall survival, in patients with clear margins after complete resection of locally advanced rectal cancer.

OUTLINE: This is an open-label, randomized, controlled, prospective, multicenter study. Patients are stratified according to surgeon and nodal status (node positive vs node negative vs unknown). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo standard follow up.
* Arm II: Patients receive oral capecitabine twice daily on days 1-14 and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 5 years, and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * Within 15 cm of the anal verge
  * Locally advanced disease
* Underwent complete resection of primary tumor within the past 12 weeks

  * ypT0-4, N0-2 with definitive histology at surgery
  * Circumferential resection margin > 1 mm
  * No gross evidence of residual disease
* Received neoadjuvant fluoropyrimidine-based chemoradiotherapy with ≥ 45 Gy planned total radiation dose, given in 1 of the following fashions:

  * Prolonged fluorouracil IV during radiotherapy
  * Low-dose leucovorin calcium and fluorouracil (days 1-5 and 29-33) concurrently with radiotherapy
  * Oral capecitabine concurrently with radiotherapy
* No evidence of metastatic disease

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine clearance ≥ 50 mL/min
* Bilirubin ≤ 1.25 times upper limit of normal (ULN)
* AST and ALT ≤ 1.25 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No known dihydropyrimidine dehydrogenase deficiency
* No hypersensitivity to platinum compounds
* No preexisting peripheral neuropathy ≥ grade 1
* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome
* No other serious uncontrolled medical condition or concurrent medical illness that would compromise life expectancy and/or preclude study compliance, including any of the following:

  * Serious uncontrolled infections
  * Significant cardiac disease (e.g., uncontrolled angina, congestive heart failure, cardiomyopathy, or arrhythmias) or myocardial infarction within the past 12 months
  * Interstitial pneumonia or symptomatic lung fibrosis
* No other malignancies except adequately treated in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin, unless disease-free for ≥ 10 years
* No history of uncontrolled seizures, CNS disorders, or psychiatric disability that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy exceeding 6 weeks in duration

  * Prior chemotherapy given as part of neoadjuvant treatment (i.e., chemoradiotherapy) may last a maximum of 11-12 weeks
* No prior oxaliplatin
* Prior mitomycin C, irinotecan hydrochloride, or cetuximab allowed
* No concurrent warfarin, antiviral agents, or phenytoin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2004-11; Primary Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Disease-free survival at 3 years

SECONDARY OUTCOMES:
Overall survival at 5 years
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Robert Glynne-Jones, MD, Study Chair — Mount Vernon Cancer Centre at Mount Vernon Hospital
Locations (72):
- United Kingdom (72):
  - Wansbeck General Hospital, Ashington, England
  - North Devon District Hospital, Barnstaple, England
  - Furness General Hospital, Barrow in Furness, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Good Hope Hospital, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Pilgrim Hospital, Boston, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Queen's Hospital, Burton-on-Trent, England
  - Cumberland Infirmary, Carlisle, England
  - Broomfield Hospital, Chelmsford, Essex, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Castle Hill Hospital, Cottingham, England
  - Walsgrave Hospital, Coventry, England
  - Derbyshire Royal Infirmary, Derby, England
  - Doncaster Royal Infirmary, Doncaster, England
  - University Hospital of North Durham, Durham, England
  - Princess Alexandra Hospital, Essex, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Royal Bolton Hospital, Farnworth, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Wycombe General Hospital, High Wycombe, England
  - Princess Royal Hospital at Hull and East Yorkshire NHS Trust, Hull, England
  - King George Hospital, Ilford, Essex, England
  - Ipswich Hospital, Ipswich, England
  - West Middlesex University Hospital, Isleworth, England
  - Kidderminster Hospital, Kidderminster Worcestershire, England
  - Royal Albert Edward Infirmary, Lancanshire, England
  - Royal Lancaster Infirmary, Lancaster, England
  - Cookridge Hospital, Leeds, England
  - Lincoln County Hospital, Lincoln, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Helen Rollason Cancer Care Centre at North Middlesex Hospital, London, England
  - Whittington Hospital, London, England
  - University College of London Hospitals, London, England
  - UCL Cancer Institute, London, England
  - St. George's Hospital, London, England
  - Charing Cross Hospital, London, England
  - Macclesfield District General Hospital, Macclesfield, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - St. Mary's Hospital, Newport, England
  - Northampton General Hospital, Northampton, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Churchill Hospital, Oxford, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Oldchurch Hospital, Romford, England
  - Hope Hospital, Salford, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Southampton General Hospital, Southampton, England
  - Southport and Formby District General Hospital, Southport, England
  - Sunderland Royal Hospital, Sunderland, England
  - Kingston Hospital, Surrey, England
  - Walsall Manor Hospital, Walsall, England
  - Sandwell General Hospital, West Bromwich, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England
  - Worcester Royal Hospital, Worcester, England
  - Yeovil District Hospital, Yeovil, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Royal Glamorgan Hospital, Lhantrisant, Wales
  - Hereford Hospitals, Hereford
  - Scarborough General Hospital, Scarborough

REFERENCES:
- [Derived] Glynne-Jones R, Counsell N, Quirke P, Mortensen N, Maraveyas A, Meadows HM, Ledermann J, Sebag-Montefiore D. Chronicle: results of a randomised phase III trial in locally advanced rectal cancer after neoadjuvant chemoradiation randomising postoperative adjuvant capecitabine plus oxaliplatin (XELOX) versus control. Ann Oncol. 2014 Jul;25(7):1356-1362. doi: 10.1093/annonc/mdu147. Epub 2014 Apr 8. PMID 24718885